CLINICAL TRIAL: NCT01354106
Title: Adhesive Tape Trauma Evaluation of Two Gentle Tapes in Healthy Human Infant Subjects
Brief Title: Adhesive Tape Trauma Evaluation of Two Gentle Tapes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EM-05-012247
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Adhesive Tape Trauma
Keywords: Skin condition after wear

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3M Kind Removal Silicone Tape (Experimental): investigational medical Silicone tape, 1" x 1.5" sample, applied on time, worn for 24 hours.
  Interventions: Device: Skin Trauma
- 3M Micropore Medical Tape (Other): Commercially available Medical Paper Tape, 1" x 1.5" sample, applied on time, worn for 24 hours. Study Control.
  Interventions: Device: Skin Trauma

INTERVENTIONS:
Device: Skin Trauma — Each participant completed received both treatment arms, the 3M Micropore and 3M Kind Removal Silicone Tape.
  Other Names: 3M Micropore; 3M Kind Removal Silicone Tape - Investigational tape

SUMMARY:
The objective of this study is to determine the relative gentleness of two tapes recognized for gentleness. A three-prong multidimensional evaluation consisting of laboratory assessments, expert skin grader and subject discomfort assessment will be used.

DETAILED DESCRIPTION:
The objective of this study is to determine the relative gentleness of a new investigational tape compared to 3M Micropore tape, a gold standard tape recognized for its gentleness and used as a mainstay in cosmetic surgery and neonatal care. A three-prong multidimensional evaluation consisting of laboratory assessments, expert skin grader and subject discomfort assessment will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Who are healthy and who have intact skin at the test site with a baseline score of 0 for erythema
2. Who are between the ages of 6 months - 4 years of age
3. Who has a Fitzpatrick Skin Type of I, II or III
4. Subject who's parent agrees to not use any products (i.e. topical medications, creams, powders or ointments) on the test sites for 24 hours prior to the study start date
5. Whose parent is willing to sign the Informed Consent Form.

Exclusion Criteria:

1. Who are known to be developmentally delayed
2. Who have sunburn, skin infection or scars, moles, or other blemishes on the back that would obscure grading of the test sites
3. Who have had any exposure to other topical medications, creams, powders, or ointments on the test sites 24 hours prior to the start of the study.
4. Who have had a strep infection within the past 2 weeks
5. Who have a history of diabetes, psoriasis, any active dermatitis, or recent history of dermatitis or skin reactions
6. Who have allergies to isocyanates, or acrylate adhesive products
7. Who currently take any antihistamines or anti-inflammatory medication or who have taken any of these medications within 48 hours prior to the start of the study or does not agree to refrain from taking these medications for the 48 hours prior to the start of the study and for the duration of the study (Tylenol is an acceptable pain reliever).

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary L Grove, PhD, Principal Investigator — cyberDERM
Locations (1):
- cyberDERM, Broomall, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment started May 16, 2011 at cyberDERM
Pre-assignment Details: participant not to use any products on the test sites for 24 hours prior to the study state date.
Groups:
- Adhesive Medical Tape: Each study participant received both treatment arms: 3M Kind Removal Silicone Tape (1" x 1.5" sample, applied one time, worn 24 hours) and 3M Micropore Silicone Tape (1" x 1.5" sample, applied one ime, worn 24 hours).
Period: Overall Study
Arm/Group | Adhesive Medical Tape
Started | 26
Completed | 24
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Infant: Investigational adhesive tape control paper tape
Arm/Group | Infant
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.88 (0.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Skin Trauma
Description: Expert grader using Erythema/Edema Scale 0=No visible response
  1. mild response
  2. moderate response
  3. severe response
  4. extreme response
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- 3M Kind Removal Silicone Tape; 3M Micropore Medical Tape: 1" x 1.5" sample applied one time, worn for 24 hours.
Arm/Group | 3M Kind Removal Silicone Tape | 3M Micropore Medical Tape
Number analyzed (Participants) | 24 | 24
Units on a scale | 0.93 (0.14) | 1.35 (0.11)

ADVERSE EVENTS:
Arm/Group | Investigational Adhesive Tape | Control Paper Tape
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The proposed disclosure must be reviewed by the sponsor. The sponsor shall complete the review within 30 working days after receipt. The PI will discuss and consider in good faith the sponsor recommendations resulting from the review.